CLINICAL TRIAL: NCT03962543
Title: A Phase 2b Trial of the MEK 1/2 Inhibitor (MEKi) PD-0325901 in Adult and Pediatric Patients With Neurofibromatosis Type 1 (NF1)-Associated Inoperable Plexiform Neurofibromas (PNs) That Are Causing Significant Morbidity
Brief Title: MEK Inhibitor Mirdametinib (PD-0325901) in Patients With Neurofibromatosis Type 1 Associated Plexiform Neurofibromas
Acronym: ReNeu
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEK-NF-201
Expanded Access: NCT05028166 (Available)
Record Dates: First submitted 2019-04-12; First posted 2019-05-24 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Plexiform Neurofibroma; Neurofibromatosis Type 1 (NF1)
Keywords: Neurofibromatosis; Neurofibromatosis 1; Plexiform Neurofibroma; PD-0325901; MEK Inhibitor; Neurofibroma; Mirdametinib
MeSH Terms: conditions — Neurofibroma, Plexiform; Neurofibromatosis 1; Neurofibromatoses; Neurofibroma | interventions — mirdametinib

STUDY DESIGN:
Intervention Model Description: All participants will receive mirdametinib (PD-0325901) at a dose of 2 mg/m^2 twice daily (maximum dose of 4 mg twice daily), calculated based on body surface area. Dose will be administered in a 3-week on, 1-week off schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mirdametinib (PD-0325901) (Experimental): Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
  Interventions: Drug: Mirdametinib (PD-0325901) oral capsule or dispersible tablet

INTERVENTIONS:
Drug: Mirdametinib (PD-0325901) oral capsule or dispersible tablet — Mirdametinib (PD-0325901) capsule or dispersible tablet
  Other Names: PD-0325901; Mirdametinib

SUMMARY:
This study evaluates mirdametinib (PD-0325901) in the treatment of symptomatic inoperable neurofibromatosis type-1 (NF1)-associated plexiform neurofibromas (PNs). All participants will receive mirdametinib (PD-0325901). Eligible participants may continue in a long-term follow-up phase.

DETAILED DESCRIPTION:
Neurofibromas are non-malignant peripheral nerve sheath tumors, which are classified as plexiform neurofibromas (PNs) if they extend longitudinally along a nerve and involve multiple fascicles. PNs are a major cause of morbidity and disfigurement in individuals with NF1, and as the tumor growth progresses, can cause a multitude of clinical problems including pain and impaired physical function. PNs have the potential to undergo malignant transformation to Malignant Peripheral Nerve Sheet Tumors (MPNST).

Mirdametinib (PD-0325901) is an orally delivered, highly selective small-molecule inhibitor of the dual specificity kinases, MEK1 and MEK2 (MAPK/ERK Kinase) which prevents the phosphorylation and subsequent activation of mitogen-activated protein kinase (MAPK).

Previous studies of mirdametinib (PD-0325901) demonstrated PN shrinkage and sustained inhibition of pERK. Reduced tumor volume indicated that cell proliferation or cell death may be altered in PNs with administration of mirdametinib (PD-0325901).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has documented NF1 mutation or a diagnosis of neurofibromatosis type 1 (NF1) using National Institute of Health (NIH) Consensus Conference criteria inclusive of the presence of a plexiform neurofibroma (PN).
* Participant has a PN that is causing significant morbidity.
* Participant has a PN that cannot be completely surgically removed.
* Participant has a target tumor that is amenable to volumetric MRI analysis.
* Participant is willing to undergo a tumor biopsy pre and post treatment if ≥ 18 years of age.
* Participant has adequate organ and bone marrow function.

Key Exclusion Criteria:

* Participant has abnormal liver function or history of liver disease.
* Participant has lymphoma, leukemia or any malignancy within the past 5 years (except for resected basal/squamous skin carcinomas without metastases within 3 years).
* Participant has breast cancer within 10 years.
* Participant has active optic glioma or other low-grade glioma requiring treatment.
* Participant has abnormal QT interval corrected or other heart disease within 6 months.
* Participant has a history of retinal pathology, risk factors for retinal vein occlusion or has a history of glaucoma.
* Participant has known malabsorption syndrome or gastrointestinal conditions that would impair absorption of mirdametinib (PD-0325901).
* Participant has received NF1 PN-targeted therapy within 45 days.
* Participant previously received or is currently receiving therapy with mirdametinib (PD-0325901) or any other MEK1/2 inhibitor.
* Participant has received radiation therapy within 6 months or has received radiation to the orbit at any time.
* Participant is unable to undergo or tolerate MRI.
* Participant has active bacterial, fungal or viral infection.
* Participant has experienced other severe acute or chronic medical or psychiatric conditions within 1 year.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2028-12-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Moertel, MD, Principal Investigator — University of Minnesota
Locations (50):
- United States (50):
  - University of Alabama at Birmingham/Children's of Alabama, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA Oncology Center, Los Angeles, California
  - University of California - Irvine Health, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - University of California - Davis Comprehensive Cancer Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours A. I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Pediatric Oncology Hematology at Orlando, Orlando, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Children's Healthcare of Atlanta - Center for Advanced Pediatrics, Atlanta, Georgia
  - University of Illinois Hospital and Health Systems, Chicago, Illinois
  - University of Chicago Medical Centers, Chicago, Illinois
  - IU Health Brain Tumor Infusion Clinic, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - University of Michigan CS Mott Children's Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine-Siteman Cancer Center, St Louis, Missouri
  - St. Joseph's Univeristy Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - UNC Medical Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Jimmy Everest Center for Cancer and Blood Disorders in Children, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Children's Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Center for Clinical and Translational Sciences, Salt Lake City, Utah
  - UVA Health, Division of Neuro-Oncology, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Swedish Medical Center - Cherry Hill Campus, Seattle, Washington
  - MACC Fund Research Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
SpringWorks Therapeutics is committed to data transparency and sharing data to further research while maintaining the privacy and confidentiality of research participants. Pertinent patient-level data from completed registrational clinical trials will be made available by SpringWorks to qualified researchers upon approval of reasonable requests following de-identification/anonymization pursuant to applicable law.

REFERENCES:
- [Derived] Moertel CL, Hirbe AC, Shuhaiber HH, Bielamowicz K, Sidhu A, Viskochil D, Weber MD, Lokku A, Smith LM, Foreman NK, Hajjar FM, McNall-Knapp RY, Weintraub L, Antony R, Franson AT, Meade J, Schiff D, Walbert T, Ambady P, Bota DA, Campen CJ, Kaur G, Klesse LJ, Maraka S, Moots PL, Nevel K, Bornhorst M, Aguilar-Bonilla A, Chagnon S, Dalvi N, Gupta P, Khatib Z, Metrock LK, Nghiemphu PL, Roberts RD, Robison NJ, Sadighi Z, Stapleton S, Babovic-Vuksanovic D, Gershon TR; ReNeu Trial Investigators; ReNeu Study Investigators. ReNeu: A Pivotal, Phase IIb Trial of Mirdametinib in Adults and Children With Symptomatic Neurofibromatosis Type 1-Associated Plexiform Neurofibroma. J Clin Oncol. 2025 Feb 20;43(6):716-729. doi: 10.1200/JCO.24.01034. Epub 2024 Nov 8. PMID 39514826

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901): Patients aged 2 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
- Treatment Phase - Adult Cohort Mirdametinib (PD-0325901): Patients aged 18 and above at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
Period: Treatment Phase
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Started | 56 | 58
Completed | 33 | 31
Not Completed | 23 | 27
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 3 | 12
Not completed — Lost to Follow-up | 1 | 2
Not completed — Radiographic PD | 9 | 3
Not completed — Participant Decision | 3 | 8
Not completed — Received procedure not compatible with MRI | 0 | 1
Not completed — Ongoing in the Treatment Phase | 4 | 0
Period: Long Term Follow-Up Phase
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Started | 28 | 26
Completed | 0 | 0
Not Completed | 28 | 26
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Radiographic PD | 1 | 0
Not completed — Sponsor Request | 1 | 0
Not completed — Participant Decision | 0 | 1
Not completed — Positive pregnancy test | 0 | 1
Not completed — Ongoing in the Long Term Follow-Up Phase Phase | 25 | 22

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (Received At Least One Dose of Mirdametinib)
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) | Total
Number analyzed (Participants) | 56 | 58 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (4.50) | 35.0 (13.17) | 22.8 (15.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 37 | 67
  Male | 26 | 21 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 9
  Not Hispanic or Latino | 44 | 52 | 96
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 5 | 16
  White | 37 | 49 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 56 | 58 | 114
Karnofsky/Lansky Score [Mean (Standard Deviation); unit: units on a scale] — Karnofsky (>= 16 years of age) and Lansky (< 16 years of age) performance scores are intended to be multiples of 10 ranging from 0 to 100 with larger scores indicating better outcomes.
  units on a scale | 94.5 (9.33) | 87.1 (7.73) | 90.7 (9.29)
Childbearing Potential at Screening [Count of Participants; unit: Participants] — Population: Based on the number of female patients in the Full Analysis Set
  Participants
    number analyzed (Participants) | 30 | 37 | 67
    Yes | 15 | 29 | 44
    No | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate at the End of the Treatment Phase.
Description: Response will be determined by a blinded centralized review of volumetric MRI. The confirmed objective response rate (complete or partial response) by the end of Treatment Phase (i.e., Cycle 24) is defined as the proportion of participants who have a confirmed ≥ 20% reduction in target tumor volume as compared to baseline as assessed by a BICR, and the response needs to be confirmed by BICR in a consecutive tumor assessment within 2 - 6 months. Partial response is defined as a ≥ 20% reduction in target tumor volume from baseline. Complete response is defined as the complete resolution of the target tumor.
Time Frame: Up to 24 months
Population: The Full Analysis Set is defined as patients who received at least one dose of Mirdametinib.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 56 | 58
percentage of patients | 51.8 [38.0 to 65.3] | 41.4 [28.6 to 55.1]

2. Secondary Outcome: Percentage of Patients With Treatment-Emergent Adverse Events.
Description: All adverse events were coded using MedDRA Version 24.0. Adverse events will be assessed according to toxicities graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Time Frame: All SAEs and AEs were collected from the time of signing ICF until 30 days after the last dose of study treatment, an average of 1 year and 10 months and up to 3 years and 10 months.
Population: The Full Analysis Set includes patients who received at least one dose of Mirdametinib.
Measure: Number; unit: percentage of patients
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 56 | 58
percentage of patients | 100 | 100

3. Secondary Outcome: Duration of Response (DOR) for Participants Who Meet Criteria for Confirmed Objective Response.
Description: Duration of response is defined as the time in months between the first instance of response that is subsequently confirmed, until the date of radiographic disease progression or death, whichever occurs first. For participants who enter the LTFU Phase, all MRI assessments in both the Treatment Phase and LTFU Phase will be used to determine duration of response. Participants without radiographic disease progression or death while on study will have their results censored to their most recent adequate (i.e. evaluable) tumor assessment date.
Time Frame: Starting on the onset of confirmed objective response in the Treatment Phase and afterwards on the 15th day of every 4 cycles (each cycle is 28 days) until disease progression or death, whichever comes first, assessed up to approximately 3 years
Population: The Full Analysis Set patients with confirmed objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 29 | 24
months | NA [NA to NA] — Not reached. Only less than 50% of the patients had events in the Pediatric cohort. | NA [NA to NA] — Not reached. Only less than 50% of the patients had events in the Adult cohort.

4. Secondary Outcome: Change From Baseline on Quality of Life (QOL) as Measured by the Pediatric Quality of Life Inventory (PedsQL) at Cycle 13, Acute Version.
Description: The PedsQL consists of a 23-item core measure of global QOL that can be completed in approximately 5 minutes. There is a total score and four subscales: physical functioning, emotional functioning, social functioning and school/work functioning. Participants ≥ 5 years of age complete an age-appropriate self-report; and parents/guardians of children ages 2-17 complete a parent proxy report of the age-specific QOL. The recall period is 7 days. PedsQL items are answered on a Likert scale with responses ranging from 0 to 4 (where 0 means it is never a problem and 4 means it is almost always a problem). These items are then reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. On this scale, higher scores indicate better outcomes. Overall scale scores are calculated as the mean of the scores for the questions in said scale (or of all questions for the total score). The change from baseline is modelled using a mixed-model for repeated measures.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set patients who are eligible for the Peds-QL assessments at baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report: Patients self-reported results aged 5 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Parent Proxy: Patients parent proxy results aged 2 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
- Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) - Self-Report: Patients self-reported results aged 18 years and above at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Parent Proxy | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) - Self-Report
Number analyzed (Participants) | 50 | 56 | 58
units on a scale
  Total Score | 4.01 [-0.74 to 8.76] | 5.64 [1.75 to 9.53] | 3.94 [0.70 to 7.17]
  School/Work Functioning | -0.02 [-7.16 to 7.13] | 1.71 [-4.02 to 7.45] | 4.67 [0.52 to 8.82]
  Social Functioning | 1.85 [-4.31 to 8.01] | 7.64 [2.91 to 12.37] | 2.28 [-1.74 to 6.29]
  Emotional Functioning | 5.60 [-0.66 to 11.86] | 8.15 [3.71 to 12.58] | 1.51 [-2.78 to 5.80]
  Physical Functioning | 6.71 [0.56 to 12.87] | 5.75 [0.35 to 11.14] | 5.90 [1.33 to 10.47]

5. Secondary Outcome: Change From Baseline in Pain as Measured by the Numeric Rating Scale-11 (NRS-11) at Cycle 13.
Description: The NRS-11 is a self-reported 11-point numerical scale that assesses pain severity. Participants ≥ 8 years of age are asked to select a number from 0 (no pain) to 10 (worst pain you can imagine) that best describes their worst pain. The recall period is 24 hours. The change from baseline is modelled using a mixed-model for repeated measures.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set patients eligible for the instrument at baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report: Patients aged 8 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
- Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) - Self-Report: Patients aged 18 and above at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) - Self-Report
Number analyzed (Participants) | 37 | 58
units on a scale | -0.79 [-1.28 to -0.29] | -1.33 [-1.83 to -0.84]

6. Secondary Outcome: Change From Baseline in Pain as Measured by the Pain Interference Index (PII) at Cycle 13.
Description: The PII assesses relevant aspects of one's life, including pain interference with activities, spending time with family/friends, mood, sleep and attention. Participants ≥ 6 years of age complete a self-report, and parents/guardians of children aged 6-17 complete a parent proxy report. The recall period is 24 hours. The PII consists of 6 questions, each asking the responder to select one number from 0 to 6 that best describes how their/their proxy's pain has impacted various items over the past 24 hours with 0 representing "Not at all" and 6 representing "Completely". The mean of the completed items is taken as the PII score for a single assessment. The PII score presented each visit will be taken as the average of the PII scores over the 7 consecutive days up to and including visit day, with no transformation applied. The change from baseline is modelled using a mixed-model for repeated measures.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set patients eligible for the instrument at baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report: Patients self-reported results aged 6 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Parent Proxy: Patients parent proxy results aged 6 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Parent Proxy | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) - Self-Report
Number analyzed (Participants) | 47 | 47 | 58
units on a scale | -0.46 [-0.83 to -0.09] | -0.26 [-0.49 to -0.03] | -0.70 [-1.02 to -0.38]

7. Other Pre Specified Outcome: Change From Baseline in Localized Strength (Dynamometer) at Cycle 13.
Description: Assessment of strength will be conducted only in the area affected by the target tumor. Measurements will be obtained using Medical Research Council (MRC) grading followed by quantitative assessments using the sponsor provided MicroFET2 dynamometer. Dynamometer assessment (in lbs) must be conducted in accordance with the study reference manual. For each participant, the sum of the dynamometer scores for the muscle groups tested will be taken as an overall score for each visit with higher scores indicating better localized strength. To assess the change from baseline at a visit, a participant will need assessments in which all the following categories, as assessed at baseline, match at that visit: side affected, position during assessment (sitting/supine/lateral decubitus), muscle group assessed. The change from baseline in localized strength measured by the sum of the dynamometer scores for the muscle groups tested will be assessed at Cycle 13.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set patients eligible for this instrument at baseline.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 15 | 23
lbs | 18.8 (31.93) | 68.5 (130.33)

8. Other Pre Specified Outcome: Change From Baseline in Range of Motion of PN-Associated Functional Impairment at Cycle 13.
Description: If motor dysfunction or weakness is evident, range of motion of the affected areas and/or joints will be measured by a goniometer.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set patients who are eligible for this instrument at baseline.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 15 | 23
degrees | -6.1 (82.06) | 17.7 (51.28)

9. Other Pre Specified Outcome: Change From Baseline in Endurance at Cycle 13.
Description: If airway or lower extremity motor dysfunction is evident, endurance will be measured by completion of a 6-minute walking test.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set patients eligible for this instrument at baseline
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 11 | 16
meters | -6.8 (60.76) | 2.2 (70.41)

10. Other Pre Specified Outcome: Time to Response Defined as the Time Between First Dose and the First Date of Objective Response That is Subsequently Confirmed.
Description: Response will be determined by a blinded centralized review of volumetric MRI. Time to response is defined as the time in months from the start of treatment to the date of first response that was subsequently confirmed.
Time Frame: Up to 24 months
Population: The Full Analysis Set patients who achieved confirmed objective response.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 29 | 24
months | 8.63 (4.801) | 9.71 (5.804)

11. Other Pre Specified Outcome: Time to Progression, From the First Dose to the First Date of a ≥ 20% Increase in Tumor Volume From Baseline.
Description: Evidence of progression or tumor growth will be determined by a blinded centralized review of volumetric MRI. Time to progression is defined as the time in months between the first treatment date until the date of radiographic disease progression. For participants who enter the LTFU Phase, all MRI assessments in both the Treatment Phase and LTFU Phase will be used to determine time to progression. Participants without radiographic disease progression will have their results censored to their most recent adequate (i.e. evaluable) tumor assessment date.
Time Frame: On the 15th day of every 4 cycles (each cycle is 28 days) until disease progression is observed, assessed up to approximately 3.5 years
Population: The Full Analysis Set defined as all patients who received at least one dose of Mirdametinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 56 | 58
months | NA [NA to NA] — NA Explanation: Not reached. Only less than 50% of the patients had events in the Pediatric cohort. | NA [NA to NA] — NA Explanation: Not reached. Only less than 50% of the patients had events in the Adult cohort.

12. Other Pre Specified Outcome: Progression Free Survival, Defined as the Time in Months From the First Dose to the Date of the First ≥ 20% Increase in Tumor Volume From Baseline or Death.
Description: Evidence of progression or tumor growth will be determined by a blinded centralized review of volumetric MRI. Progression free survival is defined as the time in months between the first treatment date, until the date of radiographic disease progression or death, whichever occurs first. For participants who enter the LTFU Phase, all MRI assessments in both the Treatment Phase and LTFU Phase will be used to determine progression free survival. Participants without radiographic disease progression or death while on study will have their results censored to their most recent adequate (i.e. evaluable) tumor assessment date.
Time Frame: On the 15th day of every 4 cycles (each cycle is 28 days) until disease progression is observed or death, whichever comes first, assessed up to approximately 3.5 years
Population: The Full Analysis Set defined as all patients who received at least one dose of Mirdametinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 56 | 58
months | NA [NA to NA] — NA Explanation: NA Explanation: Not reached. Only less than 50% of the patients had events in the Pediatric cohort. | NA [NA to NA] — NA Explanation: NA Explanation: Not reached. Only less than 50% of the patients had events in the Adult cohort.

13. Other Pre Specified Outcome: Change From Baseline in PN-Associated Disfigurement Using Standardized Photography, Centrally Reviewed.
Description: For participants with a PN that is visible and amenable to photography, changes in visible tumor aspects will be evaluated by a centralized reviewer.
Time Frame: Up to 24 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Comparison of Tumor Response to Levels of pERK and Biomarkers Indicative of Inhibition of Downstream Targets of MEK (eg, ERK Phosphorylation).
Description: Measured in tumor biopsies in participants ≥ 18 years of age.
Time Frame: Up to 24 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Acceptability of the Dispersible Tablet Formulation as Measured by the Pediatric Oral Medicine Acceptability Questionnaire (P-OMAQ)
Description: The Pediatric Oral Medicine Acceptability Questionnaire (P-OMAQ) uses a 5-point numerical rate scale to measure acceptability of use of the tablet formulation with questions related to taste, smell and administration of study medication. Participants ≥ 8 years of age complete a 12-item self-report; adult parents/caregivers responsible for oversight of study drug administration for participants ages 6 months to 17 years complete a 19-item caregiver report. Each questionnaire is provided with a "past 7 days" recall with all items using a 5-point Numerical Rate Scale (1 to 5) with higher item-scores reflecting greater oral treatment acceptability. The overall P-OMAQ-P (pediatric self-report) and P-OMAQ-C (adult caregiver) scores for a participant in the study will be taken as the mean of all answered questions on the respective questionnaire.
Time Frame: Completed only once through study completion
Population: The Full Analysis Set eligible for the instrument at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901): Patients aged 8 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
- Adult Caregiver Mirdametinib (PD-0325901): The adult caregiver of Pediatric patients aged 8 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Adult Caregiver Mirdametinib (PD-0325901)
Number analyzed (Participants) | 13 | 17
units on a scale
  P-OMAQ-P | 4.3 (0.87) | NA (NA) — Not eligible for this scale.
  P-OMAQ-C | NA (NA) — Not eligible for this scale. | 4.56 (0.586)

16. Other Pre Specified Outcome: Change From Baseline in Localized Strength (Medical Research Council (MRC) Scale Grading) at Cycle 13.
Description: If motor dysfunction or weakness is evident, strength of the affected muscle groups will be measured by dynamometer and assessed by a muscle grading scale. Medical Research Council (MRC) Scale grading (0-5) must be conducted in accordance with the study reference manual. MRC Grading is assessed on a scale of 0 to 5, with 0 representing no movement being observed, and 5 representing the muscle contracting normally against full resistance. To assess the change from baseline at a visit, a participant will need assessments in which all the following categories, as assessed at baseline, match at that visit: side affected, position during assessment (sitting/supine/lateral decubitus), muscle group assessed. The MRC Grade visit score is calculated for each participant separately, and these scores are then averaged.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set patients eligible for this instrument at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
Number analyzed (Participants) | 15 | 23
units on a scale | 0.3 (0.35) | 0.3 (0.46)

17. Other Pre Specified Outcome: Change From Baseline in Physical Function Status as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) at Cycle 13: Pediatric v2.0 Mobility 8a.
Description: PROMIS measures capability of physical functioning, with questions related to daily activities. Participants 8-17 years complete a self-report of physical function in the upper extremity or lower extremity (mobility), depending on the location of the PN. The recall period is 7 days. All PROMIS items are answered on a Likert scale with responses ranging from 1 to 5, with higher scores representing higher reported mobility. The total raw score will be calculated as the sum of the individual item responses at a given visit (total raw scale range 8-40). The total raw scores for the measure will be converted to T-scores using the applicable score conversion table in the user manual and scoring instructions (PROMIS, 2023) ranging from 14 to 59 for self-report, and 14 to 56 for parent proxy with higher scores representing higher reported mobility and better outcomes. A T-score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set eligible for the instrument at baseline.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report: Patients self-reported results aged 8 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
- Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Parent Proxy: Patients parent proxy results aged 5 to 17 years old at the time of informed consent. Mirdametinib (PD-0325901) capsule or dispersible tablet 2 mg/m^2 (maximum dose of 4 mg) by mouth twice daily
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Parent Proxy
Number analyzed (Participants) | 7 | 10
T-score | 7.0 (5.66) | 2.8 (5.67)

18. Other Pre Specified Outcome: Change From Baseline in Physical Function Status as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) at Cycle 13: Pediatric v2.0 Upper Extremities 8a.
Description: PROMIS measures capability of physical functioning, with questions related to daily activities. Participants 8-17 years complete a self-report of physical function in the upper extremity or lower extremity (mobility), depending on the location of the PN. The recall period is 7 days. All PROMIS items are answered on a Likert scale with responses ranging from 1 to 5, with higher scores representing higher physical functioning in the upper extremities. The total raw score will be calculated as the sum of the individual item responses at a given visit (total raw scale range 8-40). The total raw scores for the measure will be converted to T-scores using the applicable score conversion table in the user manual and scoring instructions (PROMIS, 2023) ranging from 10 to 57 for self-report, and 13 to 55 for parent proxy with higher scores representing higher reported physical functioning and better outcomes. A T-score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set eligible for the instrument at baseline.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Self-Report | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) - Parent Proxy
Number analyzed (Participants) | 3 | 4
T-score | 11.5 (3.54) | 9.5 (3.54)

19. Other Pre Specified Outcome: Change From Baseline in Physical Function Status as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) at Cycle 13: Adult v2.0 Physical Function 8b.
Description: PROMIS measures capability of physical functioning, with questions related to daily activities. Participants ≥ 18 years with a target PN impacting physical functioning complete a self-report of physical function. The recall period is 7 days. All PROMIS items are answered on a Likert scale with responses ranging from 1 to 5, with higher scores representing higher reported physical capability. The total raw score will be calculated as the sum of the individual item responses at a given visit (total raw scale range 8-40). The total raw scores for the measure will be converted to T-scores using the applicable score conversion table in the user manual and scoring instructions (PROMIS, 2023) ranging from 20.3 to 60.1 with higher scores representing higher reported physical functioning and better outcomes. A T-score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days), up to 12 months
Population: The Full Analysis Set eligible for the instrument at baseline.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) - Self-Report
Number analyzed (Participants) | 23
T-score | 2.42 (9.447)

ADVERSE EVENTS:
Time Frame: All SAEs and AEs were collected from the time of signing ICF until 30 days after the last dose of study treatment, an average of 1 year and 10 months and up to 3 years and 10 months.
Description: All SAEs and AEs were collected from the time of signing ICF until 30 days after the last dose of study treatment. Medical occurrences that begin before the start of study treatment but after obtaining informed consent will be recorded as AEs.
Arm/Group | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901)
All-Cause Mortality (participants affected / at risk) | 0/56 | 1/58
Serious Adverse Events (participants affected / at risk) | 8/56 | 10/58
Other Adverse Events (participants affected / at risk) | 56/56 | 57/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) (N=56) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) (N=58)
COVID-19 (Infections and infestations) | 0 | 2
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Near drowning (Injury, poisoning and procedural complications) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Device breakage (Product Issues) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase - Pediatric Cohort Mirdametinib (PD-0325901) (N=56) | Treatment Phase - Adult Cohort Mirdametinib (PD-0325901) (N=58)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 24 | 45
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 7
Rash (Skin and subcutaneous tissue disorders) | 11 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 7
Eczema (Skin and subcutaneous tissue disorders) | 8 | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 7 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 31 | 34
Nausea (Gastrointestinal disorders) | 15 | 30
Vomiting (Gastrointestinal disorders) | 22 | 22
Abdominal pain (Gastrointestinal disorders) | 15 | 10
Constipation (Gastrointestinal disorders) | 6 | 9
Abdominal pain upper (Gastrointestinal disorders) | 9 | 3
Stomatitis (Gastrointestinal disorders) | 8 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 4
Ejection fraction decreased (Investigations) | 15 | 9
SARS-CoV-2 test positive (Investigations) | 11 | 12
Blood creatine phosphokinase increased (Investigations) | 12 | 8
Weight increased (Investigations) | 9 | 4
Neutrophil count decreased (Investigations) | 7 | 0
Alanine aminotransferase increased (Investigations) | 2 | 4
Blood alkaline phosphatase increased (Investigations) | 3 | 3
White blood cell count decreased (Investigations) | 6 | 0
COVID-19 (Infections and infestations) | 14 | 13
Paronychia (Infections and infestations) | 18 | 1
Upper respiratory tract infection (Infections and infestations) | 13 | 0
Skin infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 1 | 6
Pharyngitis streptococcal (Infections and infestations) | 6 | 0
Fatigue (General disorders) | 7 | 17
Pyrexia (General disorders) | 11 | 4
Oedema peripheral (General disorders) | 2 | 6
Non-cardiac chest pain (General disorders) | 3 | 4
Headache (Nervous system disorders) | 19 | 6
Dizziness (Nervous system disorders) | 5 | 10
Paraesthesia (Nervous system disorders) | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Anxiety (Psychiatric disorders) | 2 | 6
Insomnia (Psychiatric disorders) | 4 | 3
Vision blurred (Eye disorders) | 4 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 2
Ear pain (Ear and labyrinth disorders) | 4 | 5
Hypertension (Vascular disorders) | 3 | 6
Fall (Injury, poisoning and procedural complications) | 2 | 6
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03962543/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT03962543/SAP_001.pdf